CLINICAL TRIAL: NCT00909376
Title: Is Early Second Trimester Vaginal Ultrasound Scan Associated With Adverse Perinatal Outcomes?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Dr. Ori Shen, Shaare Zedek Medical Center
Other Study IDs: 1-Ledmore
Record Dates: First submitted 2009-04-02; First posted 2009-05-28 (Estimated); Last update posted 2009-05-28 (Estimated); Status verified 2009-05

CONDITIONS: Pregnancy
Keywords: Pregnancy; Ultrasonography; outcome; adverse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 - transabdominal sonography: Women who will have a transabdominal sonography done in the early second trimester.
- 2 - transvaginal sonography: Women who will have a transvaginal sonography done in the early second trimester.

SUMMARY:
Many pregnant women have an ultrasound done of their fetus in the beginning of the second trimester of pregnancy. Some have a transvaginal sonography while others have a transabdominal one, depending on clinical parameters such as weight, scars etc. In the transvaginal ultrasound there is some amount of version of the fetus done by the examiner to maintain a better aspect of the fetus, while this is not done in a transabdominal sonography.

The objective of this trail is to determine whether having a transvaginal ultrasound as opposed to a transabdominal one has an association to adverse perinatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who choose to have a ultrasound done in the early second trimester.

Exclusion Criteria:

* More than one fetus,
* No agreement to participate in the study,
* Malformative fetus.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: pregnant women with one fetus who has no malformations.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
nuchal cord entanglement | at birth

SECONDARY OUTCOMES:
SGA | at birth
Admission to intensive care unit | at birth
meconium | at birth
fetal distress | at birth
low APGAR score | 1 minute, 5 minutes after birth
need for c section | at birth

CONTACTS AND LOCATIONS:
Overall Officials: Ori Shen, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel